CLINICAL TRIAL: NCT01242774
Title: A Phase Ib, Dose-finding Study of Oral Panobinostat (LBH589) in Combination With Idarubicin and Cytarabine Induction and High-dose Cytarabine-based Consolidation Therapy in Adult Patients Less Than or Equal to 65 Years Old With Acute Myeloid Leukemia (AML)
Brief Title: Safety & Efficacy Study of Oral Panobinostat (LBH589) With Chemotherapy in Patients < 65 Years Old With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589G2101; 2009-016809-42 (EudraCT Number)
Record Dates: First submitted 2010-10-17; First posted 2010-11-17 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2015-05

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: AML; bone marrow; abnormal blast cells of myeloid; acute leukemia; cytogenetic abnormalities; HDACi
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Chromosome Aberrations | interventions — Panobinostat

ARMS (1):
- Panobinostat (Experimental)
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Oral administration of panobinostat given 3 times a week (administered on weeks 2 and 3 of a 4 week cycle) in combination with induction chemotherapy (idarubicin and cytarabine.
  Other Names: LBH589

SUMMARY:
This study will be conducted to assess the maximum tolerated dose (MTD) of panobinostat given 3 times a week (administered on weeks 2 and 3 of a 4 week cycle) in combination with induction chemotherapy (idarubicin and cytarabine) in newly diagnosed patients with a cytopathologically confirmed diagnosis of high-risk AML, and to investigate the safety of the combination in this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed adult patients = 65 years old with a cytopathologically confirmed diagnosis of high-risk AML
* = 20% bone marrow blasts via bone marrow aspiration or biopsy
* The patient has not yet been treated for AML
* 1º or 2º AML patients with high-risk category features
* ECOG PS = 2
* Renal function and liver function limits.

Exclusion Criteria:

* Patient with a 'favorable' or 'better-risk' cytogenetic profile = t(15;17); t(8;21); or inv(16) or t(16;16)
* Patient has clinical symptoms suggestive of CNS leukemia and/or CSF findings for CNS leukemia
* Prior treatment with deacetylase inhibitors (DACi) including, panobinostat
* Impaired cardiac function
* Female patient who is pregnant or breast feeding
* Male patient who is not willing to use a barrier method of contraception

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Define the maximum tolerated dose of Panobinostat (LBH589) that can be given with standard idarubicin and ara-C chemotherapy measured by safety and tolerability. | 1 year

SECONDARY OUTCOMES:
To determine the number of patients who have safety and tolerability events | 1 year
To determine Panobinostat's pharmacokinetic parameters (study the amount of Panobinostat in a person's blood over time) following study treatments | 1 year
To determine the response of Panobinostat (LBH589) given with standard idarubicin and ara-C chemotherapy (as defined by Cheson 2003) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (5):
  - Stanford University Medical Center Stanford U, Stanford, California
  - Dana Farber Cancer Institute Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Ohio State Comprehensive Cancer Center/James Cancer Hospital Dept.ofJamesCancerHospital, Columbus, Ohio
  - Medical University of South Carolina -Hollings Cancer Center MUSC/HCC (2), Charleston, South Carolina
  - Vanderbilt University Medical Center, Clinical Trials Center Vanderbilt 3, Nashville, Tennessee
- Germany (3):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Ulm
- Spain (2):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona

REFERENCES:
- [Derived] DeAngelo DJ, Walker AR, Schlenk RF, Sierra J, Medeiros BC, Ocio EM, Rollig C, Strickland SA, Thol F, Valera SZ, Dasgupta K, Berkowitz N, Stuart RK. Safety and efficacy of oral panobinostat plus chemotherapy in patients aged 65 years or younger with high-risk acute myeloid leukemia. Leuk Res. 2019 Oct;85:106197. doi: 10.1016/j.leukres.2019.106197. Epub 2019 Aug 1. PMID 31541945
- See also: Results for CLBH589G2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13744